CLINICAL TRIAL: NCT05826470
Title: Investigator Initiated Trial to Further Evaluate the Safety and Efficacy of Trans-perineal Focal Laser Ablation of Localized Prostate Cancer Using High Frequency Micro-ultrasound Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision of the Sponsor
Sponsor: Genesis Research LLC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIO-2023-001
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; Low-risk or Favorable Intermediate Risk Prostate Cancer Who Are on an Active Surveillance Regimen
Keywords: Prostate Cancer; Laser; Focal Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser Ablation (Experimental): TRANBERG® Transperineal Micro Ultrasound guided laser ablation of Prostate Cancer.
  Interventions: Device: TRANBERG®|Thermal Therapy System

INTERVENTIONS:
Device: TRANBERG®|Thermal Therapy System — Focal laser ablation.

SUMMARY:
Trans-perineal focal laser ablation represents a promising alternative focal therapy option for patients with low-risk or favorable intermediate risk prostate cancer. FLA has been extensively utilized for over a decade in the treatment of PCa using different anatomical approaches. The proposed study differs from past ones in that a trans-perineal approach with reduced risk of infection will be used in contrast to the current trans-rectal approach. In addition, high frequency micro-ultrasound imaging will be used to enhance imaging and facilitate accurate needle placement and FLA of the index lesions.

The aim of this study is to evaluate FLA as a potential optimal therapeutic intervention based on safety, ease of use, efficacy, and cost.1 FLA holds promise for the management of localized tumors. The combination of the trans-perineal focal laser ablation and micro-ultrasound imaging will enable targeted trans-perineal fusion laser induced thermal therapy of prostate cancer lesions. This approach offers significant potential advantages over traditional interventions including:

* Improved dynamic ultrasound imaging of the lesion to be treated compared to traditional ultrasound techniques.
* Enhanced ability to visualize and spare critical structures within the prostate, including the bladder neck, neurovascular bundle (NVB), urethral sphincter and organs in close proximity including the rectum.
* Sparing these structures should translate into improved preservation of ejaculation, limited changes in sexual function and minimal transient incontinence following treatment.

DETAILED DESCRIPTION:
Device: TRANBERG® Transperineal Micro Ultrasound guided laser ablation of Prostate Cancer A perineal local anesthesia block is performed with the patient in lithotomy. The micro-ultrasound, secured to a digital stepper, is inserted and advanced. The live ultrasound image is displayed on the micro-ultrasound machine. The urologist advances the laser fiber introducer, temperature probes, and laser fiber to desired positions in the prostate using micro-ultrasound guidance. One laser fiber will be used for single or multiple treatment applications.

Target treatment is achieved once the laser applicator position is confirmed. The urologist will instruct on the desired treatment parameters to be entered into the TRANBERG® console. Real-time monitoring of the ablation zone will be done using the micro-ultrasound and temperature probes. Once the individual treatment has been completed, the applicator will be relocated to the next location, if necessary. Patients will be discharged home with instructions and contact information once stable.

Primary Outcome Measures:

The primary objective of this study is to assess the safety & tolerability of a tandem approach using micro-ultrasound imaging for FLA in patients with organ confined localized low or favorable intermediate risk Prostate Cancer.

The secondary objectives are to evaluate the efficacy of FLA in ablating the index tumor lesion, as well as clinical outcomes: erectile and sexual function as well as urinary control. In addition, volumetric changes in prostate lesions, prostate size as well as cancer control in treated areas will be assessed by both imaging (mpMRI) and pathology (prostate needle biopsy). Additional secondary objectives include:

* Determine the presence or absence of csPCa in the index lesion ablation zone (in- treatment field) at the 12 month post procedure biopsy.
* Evaluate the ability of high frequency micro-ultrasound imaging to identify the mpMRI. detected index lesion in the prostate.
* Evaluate the ability of micro-ultrasound to image the index lesion ablation size and compare ablation sizes using post procedure MRI.
* Determine the cost-benefit effectiveness of the treatment with trans-perineal focal laser ablation in office treatment under local anesthesia supplement with Nitrous Oxide sedation.
* Evaluate duration of treatment using trans-perineal focal laser ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages of 40 and 85 years
2. Ability to read, understand and agree/sign the patient informed consent in the English language.
3. Serum PSA < 20 ng/ml
4. AJCC clinical tumor stage T2b or less (according to digital rectal examination)
5. Men with localized PCa (GG 1or 2, Gleason Score 7 or less) (Low or Favorable Intermediate Risk PCa) with an MR-image detected index lesion done within three months from the time of enrollment and visible on micro-ultrasound
6. According to the decision of the investigator:

   * Patient is suitable to undergo treatment with FLA
   * Able to tolerate a procedure under local anesthesia
   * Able to undergo Nitrous Oxide sedation
   * Able to undergo MR
   * has normal rectal anatomy
7. Lesion Specificity:

   * Unilateral, with cumulative lesion volumes not comprising more than 50 percent of the lobe as determined by MRI
   * Lesion distances from the outer perimeter of the energy emitting zone of the diffuser to adjacent vital structures (bladder wall, rectal wall, neurovascular bundles, and urethra) must be ≥ 8mm
8. Minimum distance to rectal wall and other sensitive structures ≥ 8mm

Exclusion Criteria:

1. Previous prostate surgery
2. Patients with recurrent prostate cancer
3. Anticoagulant therapy
4. Gleason Grade Group 3 PCa or higher
5. Multifocal PCa other than Gleason Grade Group 1
6. Locally advanced or metastatic PCa
7. Prior or ongoing PCa treatment including surgery, radiation therapy, hormonal therapy or focal therapy
8. Previous radiation of the pelvic region
9. Intraprostatic calculus > 5mm
10. Inability to tolerate a dorsal lithotomy position under Nitrous Oxide sedation for > 90 minutes
11. ECOG Status ≥2
12. Urethral Stenosis
13. Prostate height > 5 cm anterior to posterior or a prostate volume >100 cc's

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Number of Adverse Events Related to the Treatment | 12 months
  AE and SAE will be evaluated during all visits using the CTCAE scale. Grade 3 or greater AEs based on the CTCAE v5.0 within 5 days post procedure will be considered severe and related to the study procedure.

SECONDARY OUTCOMES:
Efficacy: Extent of Tumor Ablation by Laser Application | 12 months
  To evaluate the efficacy of FLA in ablating the index tumor lesion, as well as clinical outcomes: erectile and sexual function and urinary control. Volumetric changes in prostate lesions, prostate size and cancer control in treated areas assessed by mpMRI and prostate needle biopsy. Determine the presence or absence of csPCa in the index lesion ablation zone at the 12 month post procedure biopsy. Evaluate the ability of high frequency micro-ultrasound imaging to identify the mpMRI detected index lesion in the prostate. Evaluate the ability of micro-ultrasound to image the index lesion ablation size and compare ablation sizes using post procedure MRI. Evaluate duration of treatment using trans-perineal focal laser ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Genesis Research LLC., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kayano PP, Klotz L. Current evidence for focal therapy and partial gland ablation for organ-confined prostate cancer: systematic review of literature published in the last 2 years. Curr Opin Urol. 2021 Jan;31(1):49-57. doi: 10.1097/MOU.0000000000000838. PMID 33196540